CLINICAL TRIAL: NCT02875899
Title: Surfacer System to Facilitate Access in Venous Occlusions
Acronym: SAVE
Status: Completed | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP0002
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Chronic Venous Thrombosis; Venous Thrombosis Upper Extremity; Venous Thrombosis Upper Extremity Superficial Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prospective, single-arm, multicentre, international Registry of the Surfacer System for the treatment of patients with limited or diminishing upper body venous access or pathology impeding standard access methods.The purpose of this post-market Registry is to assess the standard of care and clinical outcomes of the Surfacer System used in clinical routine according to the approved commercial indications.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter registry of the Surfacer System for patients with limited or diminishing upper body venous access or pathology impeding standard access methods. The need for long term access and lack of availability of veins has led to the development of the Surfacer System, which facilitates reliable and repeatable placement of central venous catheters and restores central venous access. Based on European legislation, this Registry is considered to be an observational study. No additional diagnostic or monitoring procedures as a result of the inclusion are applied to the patients. Available data will be collected in a protected database. Up to 30 patients will be enrolled in 5 sites in Europe. Patients requiring central venous access will be enrolled who meet inclusion and exclusion criteria and for whom the device is indicated.

ELIGIBILITY:
Inclusion Criteria: patients referred for placement of a central venous catheter

* patients with limited or diminishing upper body venous access
* pathology impeding standard access methods
* signed informed consent

Exclusion Criteria:

* vulnerable subjects or incapable of giving consent
* contraindications to central venous access based on treating physicians opinion or standard of care
* occlusion of the right femoral vein
* occlusion of the iliac vein
* occlusion of the inferior vena
* acute thrombosis within a vessel (IVC, brachiocephalic and subclavian)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients requiring central venous access for:
  * dialysis
  * chemotherapy nutrition
  * delivery of any pharmacological therapy
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Absence of all acute safety and device related serious adverse event recorded on case report forms | Procedure through discharge at 24 hours post procedure. Data will be presented through study completion, 1 year.
  overall complication rate compared to safety data

SECONDARY OUTCOMES:
Ability to place central venous access catheter using Surfacer system | Procedure
  performance evaluated by procedure time measured by time to create access
Surfacer system advancement of the exit wire outside the vein | procedure
  Ability to advance system from femoral vein to supraclavicular exit as measured by time
Insertion of a standard central venous access catheter to deliver fluid or pharmacological agents | procedure
  introducing a standard central venous access catheter over the needle wire

CONTACTS AND LOCATIONS:
Overall Officials: Laura Minarsch, RT, Study Director — Bluegrass Vascular
Locations (4):
- University of Vienna, Vienna, Waehringer Guertel 18-20, Austria
- Germany (2):
  - University Hospital of Cologne, Cologne
  - Schon Klinik, Düsseldorf
- Azienda Ospedaliera San Carlo Borromeo, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elayi CS, Allen CL, Leung S, Lusher S, Morales GX, Wiisanen M, Aikat S, Kakavand B, Shah JS, Moliterno DJ, Gurley JC. Inside-out access: a new method of lead placement for patients with central venous occlusions. Heart Rhythm. 2011 Jun;8(6):851-7. doi: 10.1016/j.hrthm.2011.01.024. Epub 2011 Jan 13. PMID 21237290
- [Background] Frykholm P, Pikwer A, Hammarskjold F, Larsson AT, Lindgren S, Lindwall R, Taxbro K, Oberg F, Acosta S, Akeson J. Clinical guidelines on central venous catheterisation. Swedish Society of Anaesthesiology and Intensive Care Medicine. Acta Anaesthesiol Scand. 2014 May;58(5):508-24. doi: 10.1111/aas.12295. Epub 2014 Mar 5. PMID 24593804
- [Background] Baskin JL, Pui CH, Reiss U, Wilimas JA, Metzger ML, Ribeiro RC, Howard SC. Management of occlusion and thrombosis associated with long-term indwelling central venous catheters. Lancet. 2009 Jul 11;374(9684):159-69. doi: 10.1016/S0140-6736(09)60220-8. PMID 19595350